CLINICAL TRIAL: NCT04884776
Title: Modulation of Gut Microbiota to Enhance Health and Immunity of Vulnerable Individuals During COVID-19 Pandemic
Brief Title: Modulation of Gut Microbiota to Enhance Health and Immunity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Mak Wing Yan, Assistant Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IMPACT Study
Record Dates: First submitted 2021-04-29; First posted 2021-05-13 (Actual); Last update posted 2022-12-29 (Actual); Status verified 2022-12

CONDITIONS: Gut Microbiota; COVID-19 Vaccine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active arm (Active Comparator): Subject will be instructed to take microbiome immunity formula 2 sachets daily for a total of 12 weeks.
  Interventions: Dietary Supplement: Microbiome immunity formula
- Placebo arm (Placebo Comparator): Subject will be instructed to take active placebo daily for a total of 12 weeks.
  Interventions: Dietary Supplement: Active placebo

INTERVENTIONS:
Dietary Supplement: Microbiome immunity formula — Microbiome immunity formula contains probiotics blend (3 Bifidobacteria, 10 billion CFU per sachet)
  Arms: Active arm
Dietary Supplement: Active placebo — Active placebo contains active vitamin
  Arms: Placebo arm

SUMMARY:
The novel coronavirus infection (COVID-19) caused by the SARS-CoV-2 virus is now a pandemic and has culminated major morbidity and mortality globally. Studies have shown that patients with underlying type 2 diabetes mellitus (DM), obesity, old age and hypertension had a higher risk of developing severe COVID-19 infection and mortality related to COVID-19.Emerging evidence has shown that gut microbiota plays an important role in the pathogenesis of COVID-19.

DETAILED DESCRIPTION:
HYPOTHESIS We hypothesize that modulating the gut microbiota with a microbiome immunity formula can rebalance the gut microbiota in populations at risk of infection, like, patients with type 2 DM and elderlies and can lower the number of hospitalisation and reduce side effects associated with COVID-19 vaccination.

AIM We aim to evaluate the efficacy of modulating gut microbiota with a microbiome immunity formula in vulnerable subjects (patients with underlying type 2 DM and elderlies) in improving immune functions, reducing adverse events associated with COVID-19 vaccinations and reducing hospitalisation in susceptible individuals during the COVID-19 pandemic.

STUDY DESIGN This is a double-blinded, randomized, active-placebo controlled study comparing a microbiome immunity formula and placebo in enhancing immunity and reducing hospitalisation within one year. Except two kinds of subjects (Substudy 1: Patients with Type 2 DM and Substudy 2: Elderly individual) will be included in respective substudy, all other methodologies are the same. In each substudy, at least half of the recruited subjects will plan to receive COVID-19 vaccination and start to take the study products after vaccination. Recruited subjects will be randomised to receive a microbiome immunity formula or active placebo for 3 months, with another 9 months follow-up after completion of study products.

ELIGIBILITY:
Substudy 1

Inclusion Criteria:

1. Age 18 years - below 65 years
2. A confirmed diagnosis of type 2 DM for ≥ 3 months with stable control (i.e. no change in DM medications in recent 2 months)
3. Written informed consents obtained

Exclusion Criteria:

1. Known history of confirmed COVID-19 infection
2. Known active sepsis or active malignancy
3. Known increased infection risk due to underlying immunosuppressed state which includes:

   * Prior organ or hematopoietic stem cell transplant
   * Neutropenia with absolute neutrophil count (ANC) <500 cells/ul at the time of study inclusion
   * Known HIV infection with CD4 <200 cells/ul at the time of study inclusion
   * On concomitant immunosuppressants or corticosteroid at a dose of prednisolone equivalent dose 10mg or more for more than 3 months
4. Known history or active infective endocarditis
5. On peritoneal dialysis or haemodialysis
6. Documented pregnancy

Substudy 2

Inclusion Criteria:

1. Age 65 years and above
2. Written informed consents obtained

Exclusion Criteria:

1. Known history of confirmed COVID-19 infection
2. Known active sepsis or active malignancy
3. Known increased infection risk due to underlying immunosuppressed state which includes:

   * Prior organ or hematopoietic stem cell transplant
   * Neutropenia with absolute neutrophil count (ANC) <500 cells/ul at the time of study inclusion
   * Known HIV infection with CD4 <200 cells/ul at the time of study inclusion
   * On concomitant immunosuppressants, chemotherapies or corticosteroid at a dose of prednisolone equivalent dose 10mg or more for more than 3 months
4. Known history or active infective endocarditis
5. On peritoneal dialysis or haemodialysis
6. Known active malignancy
7. Known terminal illness with life expectancy less than 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 453 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2024-05-31 (Estimated); Study Completion 2024-05-31 (Estimated)

PRIMARY OUTCOMES:
Adverse events/Serious adverse events | within 6 months
  Proportion of patients who presented with new symptoms/diseases which exerted unfavourable impacts on subjects. Serious adverse events are those adverse clinical events that resulted in hospital admission and/or death

SECONDARY OUTCOMES:
Immunogenicity of the COVID-19 vaccine | 3 months and 6 months
  Measured by serum neutralization assay against pseudo virus and live virus, and IgM and IgG against receptor-binding domain [RBD] and S1
Change in gut microbiome | 1, 3, 6, and 12 months
  Measured the gut microbiome changes by metagenomic sequencing and metabolite profiling by targeted and/or untargeted metabolites profiling
Changes in plasma inflammatory cytokines | 3 months and 6 months
  Measured the inflammatory cytokines (CRP or ESR) in blood result
Restoration of gut dysbiosis | 1, 3, 6 and 12 months
  It is defined as improvement in (i) gut microbiome composition and diversity; (ii) functional potential (i.e., MetaCyc pathway abundances); and (iii) proliferation of beneficial bacteria genus (i.e., bifidobacteria, eubacterium, roseburia and other short-chain fatty acids producers
Number of unscheduled hospitalisation and clinic visits | 1, 3, 6, and 12 months
  Number of unscheduled hospitalisation and clinic visits
Changes of quality of life | 1, 3, 6, and 12 months
  Measured the score of EQ-5D-5L which measure the health-related quality of life
Changes in glycaemic control | 1, 6 and 12 months
  Measured by HbA1c

CONTACTS AND LOCATIONS:
Overall Officials: Joyce WY Mak, FHKAM, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Shatin, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhou F, Yu T, Du R, Fan G, Liu Y, Liu Z, Xiang J, Wang Y, Song B, Gu X, Guan L, Wei Y, Li H, Wu X, Xu J, Tu S, Zhang Y, Chen H, Cao B. Clinical course and risk factors for mortality of adult inpatients with COVID-19 in Wuhan, China: a retrospective cohort study. Lancet. 2020 Mar 28;395(10229):1054-1062. doi: 10.1016/S0140-6736(20)30566-3. Epub 2020 Mar 11. PMID 32171076
- [Background] McGurnaghan SJ, Weir A, Bishop J, Kennedy S, Blackbourn LAK, McAllister DA, Hutchinson S, Caparrotta TM, Mellor J, Jeyam A, O'Reilly JE, Wild SH, Hatam S, Hohn A, Colombo M, Robertson C, Lone N, Murray J, Butterly E, Petrie J, Kennon B, McCrimmon R, Lindsay R, Pearson E, Sattar N, McKnight J, Philip S, Collier A, McMenamin J, Smith-Palmer A, Goldberg D, McKeigue PM, Colhoun HM; Public Health Scotland COVID-19 Health Protection Study Group; Scottish Diabetes Research Network Epidemiology Group. Risks of and risk factors for COVID-19 disease in people with diabetes: a cohort study of the total population of Scotland. Lancet Diabetes Endocrinol. 2021 Feb;9(2):82-93. doi: 10.1016/S2213-8587(20)30405-8. Epub 2020 Dec 23. PMID 33357491
- [Background] Richardson S, Hirsch JS, Narasimhan M, Crawford JM, McGinn T, Davidson KW; the Northwell COVID-19 Research Consortium; Barnaby DP, Becker LB, Chelico JD, Cohen SL, Cookingham J, Coppa K, Diefenbach MA, Dominello AJ, Duer-Hefele J, Falzon L, Gitlin J, Hajizadeh N, Harvin TG, Hirschwerk DA, Kim EJ, Kozel ZM, Marrast LM, Mogavero JN, Osorio GA, Qiu M, Zanos TP. Presenting Characteristics, Comorbidities, and Outcomes Among 5700 Patients Hospitalized With COVID-19 in the New York City Area. JAMA. 2020 May 26;323(20):2052-2059. doi: 10.1001/jama.2020.6775. PMID 32320003
- [Background] Grasselli G, Zangrillo A, Zanella A, Antonelli M, Cabrini L, Castelli A, Cereda D, Coluccello A, Foti G, Fumagalli R, Iotti G, Latronico N, Lorini L, Merler S, Natalini G, Piatti A, Ranieri MV, Scandroglio AM, Storti E, Cecconi M, Pesenti A; COVID-19 Lombardy ICU Network. Baseline Characteristics and Outcomes of 1591 Patients Infected With SARS-CoV-2 Admitted to ICUs of the Lombardy Region, Italy. JAMA. 2020 Apr 28;323(16):1574-1581. doi: 10.1001/jama.2020.5394. PMID 32250385
- [Background] Apicella M, Campopiano MC, Mantuano M, Mazoni L, Coppelli A, Del Prato S. COVID-19 in people with diabetes: understanding the reasons for worse outcomes. Lancet Diabetes Endocrinol. 2020 Sep;8(9):782-792. doi: 10.1016/S2213-8587(20)30238-2. Epub 2020 Jul 17. PMID 32687793
- [Background] Quan J, Li TK, Pang H, Choi CH, Siu SC, Tang SY, Wat NMS, Woo J, Johnston JM, Leung GM. Diabetes incidence and prevalence in Hong Kong, China during 2006-2014. Diabet Med. 2017 Jul;34(7):902-908. doi: 10.1111/dme.13284. Epub 2016 Nov 29. PMID 27859570
- [Background] Mueller AL, McNamara MS, Sinclair DA. Why does COVID-19 disproportionately affect older people? Aging (Albany NY). 2020 May 29;12(10):9959-9981. doi: 10.18632/aging.103344. Epub 2020 May 29. PMID 32470948
- [Background] Marquez EJ, Chung CH, Marches R, Rossi RJ, Nehar-Belaid D, Eroglu A, Mellert DJ, Kuchel GA, Banchereau J, Ucar D. Sexual-dimorphism in human immune system aging. Nat Commun. 2020 Feb 6;11(1):751. doi: 10.1038/s41467-020-14396-9. PMID 32029736
- [Background] Jaillon S, Berthenet K, Garlanda C. Sexual Dimorphism in Innate Immunity. Clin Rev Allergy Immunol. 2019 Jun;56(3):308-321. doi: 10.1007/s12016-017-8648-x. PMID 28963611
- [Background] Yeoh YK, Zuo T, Lui GC, Zhang F, Liu Q, Li AY, Chung AC, Cheung CP, Tso EY, Fung KS, Chan V, Ling L, Joynt G, Hui DS, Chow KM, Ng SSS, Li TC, Ng RW, Yip TC, Wong GL, Chan FK, Wong CK, Chan PK, Ng SC. Gut microbiota composition reflects disease severity and dysfunctional immune responses in patients with COVID-19. Gut. 2021 Apr;70(4):698-706. doi: 10.1136/gutjnl-2020-323020. Epub 2021 Jan 11. PMID 33431578
- [Background] Segal JP, Mak JWY, Mullish BH, Alexander JL, Ng SC, Marchesi JR. The gut microbiome: an under-recognised contributor to the COVID-19 pandemic? Therap Adv Gastroenterol. 2020 Nov 24;13:1756284820974914. doi: 10.1177/1756284820974914. eCollection 2020. PMID 33281941
- [Background] Zhang X, Tan Y, Ling Y, Lu G, Liu F, Yi Z, Jia X, Wu M, Shi B, Xu S, Chen J, Wang W, Chen B, Jiang L, Yu S, Lu J, Wang J, Xu M, Yuan Z, Zhang Q, Zhang X, Zhao G, Wang S, Chen S, Lu H. Viral and host factors related to the clinical outcome of COVID-19. Nature. 2020 Jul;583(7816):437-440. doi: 10.1038/s41586-020-2355-0. Epub 2020 May 20. PMID 32434211
- [Background] Zuo T, Zhang F, Lui GCY, Yeoh YK, Li AYL, Zhan H, Wan Y, Chung ACK, Cheung CP, Chen N, Lai CKC, Chen Z, Tso EYK, Fung KSC, Chan V, Ling L, Joynt G, Hui DSC, Chan FKL, Chan PKS, Ng SC. Alterations in Gut Microbiota of Patients With COVID-19 During Time of Hospitalization. Gastroenterology. 2020 Sep;159(3):944-955.e8. doi: 10.1053/j.gastro.2020.05.048. Epub 2020 May 20. PMID 32442562
- [Background] Zuo T, Liu Q, Zhang F, Lui GC, Tso EY, Yeoh YK, Chen Z, Boon SS, Chan FK, Chan PK, Ng SC. Depicting SARS-CoV-2 faecal viral activity in association with gut microbiota composition in patients with COVID-19. Gut. 2021 Feb;70(2):276-284. doi: 10.1136/gutjnl-2020-322294. Epub 2020 Jul 20. PMID 32690600
- [Background] Belkaid Y, Hand TW. Role of the microbiota in immunity and inflammation. Cell. 2014 Mar 27;157(1):121-41. doi: 10.1016/j.cell.2014.03.011. PMID 24679531
- [Background] Takiishi T, Fenero CIM, Camara NOS. Intestinal barrier and gut microbiota: Shaping our immune responses throughout life. Tissue Barriers. 2017 Oct 2;5(4):e1373208. doi: 10.1080/21688370.2017.1373208. Epub 2017 Sep 28. PMID 28956703
- [Background] Levy M, Kolodziejczyk AA, Thaiss CA, Elinav E. Dysbiosis and the immune system. Nat Rev Immunol. 2017 Apr;17(4):219-232. doi: 10.1038/nri.2017.7. Epub 2017 Mar 6. PMID 28260787
- [Background] Qin J, Li Y, Cai Z, Li S, Zhu J, Zhang F, Liang S, Zhang W, Guan Y, Shen D, Peng Y, Zhang D, Jie Z, Wu W, Qin Y, Xue W, Li J, Han L, Lu D, Wu P, Dai Y, Sun X, Li Z, Tang A, Zhong S, Li X, Chen W, Xu R, Wang M, Feng Q, Gong M, Yu J, Zhang Y, Zhang M, Hansen T, Sanchez G, Raes J, Falony G, Okuda S, Almeida M, LeChatelier E, Renault P, Pons N, Batto JM, Zhang Z, Chen H, Yang R, Zheng W, Li S, Yang H, Wang J, Ehrlich SD, Nielsen R, Pedersen O, Kristiansen K, Wang J. A metagenome-wide association study of gut microbiota in type 2 diabetes. Nature. 2012 Oct 4;490(7418):55-60. doi: 10.1038/nature11450. Epub 2012 Sep 26. PMID 23023125
- [Background] Stenman LK, Waget A, Garret C, Briand F, Burcelin R, Sulpice T, Lahtinen S. Probiotic B420 and prebiotic polydextrose improve efficacy of antidiabetic drugs in mice. Diabetol Metab Syndr. 2015 Sep 12;7:75. doi: 10.1186/s13098-015-0075-7. eCollection 2015. PMID 26366205
- [Background] Reimer RA, Grover GJ, Koetzner L, Gahler RJ, Lyon MR, Wood S. Combining sitagliptin/metformin with a functional fiber delays diabetes progression in Zucker rats. J Endocrinol. 2014 Feb 10;220(3):361-73. doi: 10.1530/JOE-13-0484. Print 2014 Mar. PMID 24389593
- [Background] Zheng J, Li H, Zhang X, Jiang M, Luo C, Lu Z, Xu Z, Shi J. Prebiotic Mannan-Oligosaccharides Augment the Hypoglycemic Effects of Metformin in Correlation with Modulating Gut Microbiota. J Agric Food Chem. 2018 Jun 13;66(23):5821-5831. doi: 10.1021/acs.jafc.8b00829. Epub 2018 Jun 5. PMID 29701959
- [Background] Landete JM, Gaya P, Rodriguez E, Langa S, Peiroten A, Medina M, Arques JL. Probiotic Bacteria for Healthier Aging: Immunomodulation and Metabolism of Phytoestrogens. Biomed Res Int. 2017;2017:5939818. doi: 10.1155/2017/5939818. Epub 2017 Oct 1. PMID 29109959
- [Background] Peterson CT, Sharma V, Elmen L, Peterson SN. Immune homeostasis, dysbiosis and therapeutic modulation of the gut microbiota. Clin Exp Immunol. 2015 Mar;179(3):363-77. doi: 10.1111/cei.12474. PMID 25345825
- [Background] Yan F, Polk DB. Probiotics and immune health. Curr Opin Gastroenterol. 2011 Oct;27(6):496-501. doi: 10.1097/MOG.0b013e32834baa4d. PMID 21897224
- [Background] Maldonado Galdeano C, Cazorla SI, Lemme Dumit JM, Velez E, Perdigon G. Beneficial Effects of Probiotic Consumption on the Immune System. Ann Nutr Metab. 2019;74(2):115-124. doi: 10.1159/000496426. Epub 2019 Jan 23. PMID 30673668
- [Background] de Jong SE, Olin A, Pulendran B. The Impact of the Microbiome on Immunity to Vaccination in Humans. Cell Host Microbe. 2020 Aug 12;28(2):169-179. doi: 10.1016/j.chom.2020.06.014. PMID 32791110
- [Background] Hagan T, Cortese M, Rouphael N, Boudreau C, Linde C, Maddur MS, Das J, Wang H, Guthmiller J, Zheng NY, Huang M, Uphadhyay AA, Gardinassi L, Petitdemange C, McCullough MP, Johnson SJ, Gill K, Cervasi B, Zou J, Bretin A, Hahn M, Gewirtz AT, Bosinger SE, Wilson PC, Li S, Alter G, Khurana S, Golding H, Pulendran B. Antibiotics-Driven Gut Microbiome Perturbation Alters Immunity to Vaccines in Humans. Cell. 2019 Sep 5;178(6):1313-1328.e13. doi: 10.1016/j.cell.2019.08.010. PMID 31491384
- [Background] Davidson LE, Fiorino AM, Snydman DR, Hibberd PL. Lactobacillus GG as an immune adjuvant for live-attenuated influenza vaccine in healthy adults: a randomized double-blind placebo-controlled trial. Eur J Clin Nutr. 2011 Apr;65(4):501-7. doi: 10.1038/ejcn.2010.289. Epub 2011 Feb 2. PMID 21285968
- [Background] Torjesen I. Covid-19: Norway investigates 23 deaths in frail elderly patients after vaccination. BMJ. 2021 Jan 15;372:n149. doi: 10.1136/bmj.n149. No abstract available. PMID 33451975